CLINICAL TRIAL: NCT01349660
Title: Phase I/II Study of the Combination of BKM120 and Bevacizumab in Patients With Refractory Solid Tumors (Phase I) and Relapsed/Refractory Glioblastoma Multiforme (Phase II)
Brief Title: Combination of BKM120 and Bevacizumab in Refractory Solid Tumors and Relapsed/Refractory Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI CNS 13
Record Dates: First submitted 2011-04-25; First posted 2011-05-06 (Estimated); Results first posted 2018-01-31 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma multiforme; GBM; Bevacizumab; PI3K Pathway; BKM120
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BKM120/Bevacizumab (Experimental): Phase I:
  BKM 120 orally (PO) once daily (dose is 60mg or 80mg). Bevacizumab: 10mg/kg intravenous (IV) every 2 weeks
  Phase II:
  BKM 120 orally (PO) once daily - dose is optimal dose determined in Phase I. Bevacizumab: 10mg/kg intravenous (IV) every 2 weeks
  Interventions: Drug: Bevacizumab; Drug: BKM120

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 10 mg/kg IV every 2 weeks
  Other Names: Avastin
Drug: BKM120 — BKM120 orally (PO) once daily
  Other Names: Buparlisib

SUMMARY:
In this phase I/II study,investigators are evaluating the feasibility and efficacy of the combination of BKM120, an oral inhibitor of PI3 kinase, and bevacizumab in the treatment of patients with relapsed/refractory GBM. In the Phase I part of the trial, the optimal BKM120 dose to be administered with a standard dose of bevacizumab will be determined in patients with refractory solid tumors. Although it is unlikely that the concurrent administration of bevacizumab will alter the pharmacokinetics of BKM120, limited pharmacokinetic sampling will be performed on all patients treated during the Phase II portion of the study. Assuming this combination is feasible, the Phase II portion of the study will proceed, using the doses determined in the Phase I portion. In the phase II portion, eligible patients will be limited to those with recurrent/progressive GBM following 1st line combined modality therapy.

DETAILED DESCRIPTION:
This is an open-label, non-randomized Phase I study of patients with advanced refractory solid tumors followed by a Phase II study for the second-line treatment of patients with relapsed/refractory glioblastoma multiforme.

In the phase I part of the study the optimal dose of BKM120 when combined with bevacizumab was determined. In the Phase II part of this study, patients with relapsed/refractory GBM following first line therapy are being treated with the BKM120/bevacizumab combination. Limited BKM120 pharmacokinetic evaluation will be performed on all patients treated during this part of the study. Patients will be reevaluated for response to treatment after 2 cycles (8 weeks). Patients with objective response or stable disease will continue treatment, with subsequent reevaluations every 8 weeks, until disease progression or unacceptable toxicity occurs.

Two populations of patients with relapsed/refractory GBM will be treated in the Phase II trial: 1) patients with no previous exposure to bevacizumab (N= 55) and 2) patients who received bevacizumab as part of first-line combined modality treatment (N= 20).

ELIGIBILITY:
Inclusion Criteria:

Phase I ONLY:

* Advanced, metastatic solid tumor that has progressed after standard therapy, or is a tumor type resistant to therapy, and for which bevacizumab is clinically appropriate.
* Patient may have measurable disease or non-measureable disease as defined by RECIST v1.1 criteria

Phase II ONLY:

* Progressive GBM after treatment with surgical resection (if possible) and 1st line radiation/chemotherapy.
* No previous treatment with a PI3K inhibitor. Previous treatment with bevacizumab as a component of first-line therapy is allowed.
* At least one measurable or evaluable lesion definable by MRI scan. Disease must be measurable by RANO criteria.
* Archival tumor tissue available for correlative testing.

ALL PATIENTS:

* Patient must be ≥ 4 weeks from administration of last dose of cancer therapy (including radiation therapy, biologic therapy, hormonal therapy, or chemotherapy). Patients who receive a small molecule targeted therapy as part of their first line treatment regimen must be ≥ 4 weeks or ≥ 5 half lives from administration of last dose, whichever is shorter. The patient must have recovered from or come to a new chronic or stable baseline from all treatment-related toxicities.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Life expectancy of ≥ 3 months.
* Adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

* Patients with diarrhea ≥ grade 2.
* Patients with uncontrolled type I or type II diabetes mellitus, defined as a fasting plasma glucose ≥120 mg/dL.
* Patients who have received prior treatment with a P13K inhibitor.
* Treatment with therapeutic doses of coumarin-type anticoagulants (maximum daily dose of 1 mg allowed for port line patency permitted).
* Patient has active cardiac disease including any of the following:

  * Left ventricular ejection fraction (LVEF) < 50% as determined by Multiple Grated acquisition (MUGA) scan or echocardiogram (ECHO)
  * QTc > 480 msec on screening ECG (using the QTcF formula)
  * Angina pectoris that requires the use of anti-anginal medication
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  * Conduction abnormality requiring a pacemaker
  * Valvular disease with documented compromise in cardiac function
  * Symptomatic pericarditis
* Patients who are currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug.
* Patients with clinical history of hemoptysis or hematemesis (defined as having bright red blood of ½ teaspoon or more per episode) ≤1 month prior to study enrollment.
* Patients with any history of a bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* Patients who have received chemotherapy or targeted anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug must recover to a grade 1 before starting the trial.
* Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) ≤ 5 effective half lives prior to starting study drug or who have not recovered from side effects of such therapy.
* Patients who have been treated with any hematopoietic colony-stimulating factors (e.g. G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment may be continued.
* Major surgical procedure, open biopsy, intracranial biopsy, ventriculoperitoneal shunt or significant traumatic injury ≤ 28 days prior to entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-12; Primary Completion 2016-12 (Actual); Study Completion 2018-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent Shih, MD, Study Chair — Sarah Cannon
Locations (8):
- United States (8):
  - Yale School of Medicine, New Haven, Connecticut
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Grand Rapids Oncology Program, Grand Rapids, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Tennessee Oncology, Nashville, Tennessee

REFERENCES:
- [Background] Bleehen NM, Stenning SP. A Medical Research Council trial of two radiotherapy doses in the treatment of grades 3 and 4 astrocytoma. The Medical Research Council Brain Tumour Working Party. Br J Cancer. 1991 Oct;64(4):769-74. doi: 10.1038/bjc.1991.396. PMID 1654987
- [Background] Bokstein F, Shpigel S, Blumenthal DT. Treatment with bevacizumab and irinotecan for recurrent high-grade glial tumors. Cancer. 2008 May 15;112(10):2267-73. doi: 10.1002/cncr.23401. PMID 18327820
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Vredenburgh JJ, Desjardins A, Herndon JE 2nd, Marcello J, Reardon DA, Quinn JA, Rich JN, Sathornsumetee S, Gururangan S, Sampson J, Wagner M, Bailey L, Bigner DD, Friedman AH, Friedman HS. Bevacizumab plus irinotecan in recurrent glioblastoma multiforme. J Clin Oncol. 2007 Oct 20;25(30):4722-9. doi: 10.1200/JCO.2007.12.2440. PMID 17947719
- [Background] Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorensen AG, Galanis E, Degroot J, Wick W, Gilbert MR, Lassman AB, Tsien C, Mikkelsen T, Wong ET, Chamberlain MC, Stupp R, Lamborn KR, Vogelbaum MA, van den Bent MJ, Chang SM. Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group. J Clin Oncol. 2010 Apr 10;28(11):1963-72. doi: 10.1200/JCO.2009.26.3541. Epub 2010 Mar 15. PMID 20231676
- [Background] Macdonald DR, Cascino TL, Schold SC Jr, Cairncross JG. Response criteria for phase II studies of supratentorial malignant glioma. J Clin Oncol. 1990 Jul;8(7):1277-80. doi: 10.1200/JCO.1990.8.7.1277. PMID 2358840
- [Background] Chakravarti A, Zhai G, Suzuki Y, Sarkesh S, Black PM, Muzikansky A, Loeffler JS. The prognostic significance of phosphatidylinositol 3-kinase pathway activation in human gliomas. J Clin Oncol. 2004 May 15;22(10):1926-33. doi: 10.1200/JCO.2004.07.193. PMID 15143086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between Oct 2011 and May 2012, 12 participants with refractory solid tumors were enrolled into the Phase I dose escalation trial from 3 U.S. investigational sites. Once a maximum tolerated dose was assigned, from Jul 2012 to Jun 2016, 76 patients with glioblastoma multiforme were enrolled in the Phase II trial from 7 U.S investigational sites
Groups:
- Phase I - Dose Level 1 (60 mg BKM, 10mg/kg Bevacizumab): BKM120: 60mg by mouth (PO), once a day for each 28 day cycle. Bevacizumab: 10 mg/kg administered intravenously (IV) on Day 1 and Day 15 of each 28 day cycle
  Phase I patients include those diagnosed with advanced, metastatic solid tumors.
- Phase I - Dose Level 2 (80 mg BKM120, 10mg/kg Bevacizumab): BKM120: 80mg by mouth (PO), once a day for each 28 day cycle. Bevacizumab: 10 mg/kg administered intravenously (IV) on Day 1 and Day 15 of each 28 day cycle.
  Phase I patients include those diagnosed with advanced, metastatic solid tumors.
- Phase II - (60 mg BKM120, 10mg/kg Bevacizumab): BKM120: 60mg by mouth (PO), once a day for each 28 day cycle. Bevacizumab: 10 mg/kg administered intravenously (IV) on Day 1 and Day 15 of each 28 day cycle.
  Phase II patients include those with progressive glioblastoma multiforme
Period: Overall Study
Arm/Group | Phase I - Dose Level 1 (60 mg BKM, 10mg/kg Bevacizumab) | Phase I - Dose Level 2 (80 mg BKM120, 10mg/kg Bevacizumab) | Phase II - (60 mg BKM120, 10mg/kg Bevacizumab)
Started | 6 | 6 | 76
Completed | 0 | 0 | 0
Not Completed | 6 | 6 | 76
Not completed — Still Receiving Study Treatment | 0 | 0 | 1
Not completed — Disease Progression | 2 | 4 | 50
Not completed — Adverse Event | 1 | 1 | 12
Not completed — Withdrawal by Subject | 2 | 0 | 9
Not completed — Death | 1 | 1 | 0
Not completed — Non-Permitted Interventions | 0 | 0 | 2
Not completed — Study Compliance | 0 | 0 | 1
Not completed — Declining Performance Status | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients that received at least one dose of study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I - Dose Level 1 (60 mg BKM, 10mg/kg Bevacizumab) | Phase I - Dose Level 2 (80 mg BKM120, 10mg/kg Bevacizumab) | Phase II - (60 mg BKM120, 10mg/kg Bevacizumab) | Total
Number analyzed (Participants) | 6 | 6 | 76 | 88
Age, Continuous [Median (Full Range); unit: years] | 61 [44 to 82] | 64 [43 to 82] | 57 [19 to 77] | 57 [19 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 36 | 40
  Male | 4 | 4 | 40 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 5 | 5
  White | 6 | 6 | 70 | 82
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 76 | 88
Primary Tumor Type [Count of Participants; unit: Participants]
  Glioblastoma Multiforme | 2 | 3 | 76 | 81
  Colorectal | 2 | 3 | 0 | 5
  Lung | 2 | 0 | 0 | 2
Prior Treatment with Bevacizumab [Count of Participants; unit: Participants] — Population: Phase I Outcomes do not utilize prior bevacizumab treatment status, thus number of participants with prior bevacizumab treatment not reported.
  Participants
    number analyzed (Participants) | 0 | 0 | 76 | 76
    Prior Bevacizumab Treatment |  |  | 19 | 19
    Bevacizumab Naive |  |  | 57 | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Phase I Patients Receiving 60mg or 80mg BKM120 Experiencing a Dose-Limiting Toxicity (DLT) to Determine the Optimal Dosage
Description: The optimal dose of BKM120 to administer in combination with standard dose bevacizumab determined as the dose at which ≤1 of 6 patients experiences a DLT assessed using NCI CTCAE v4.03 during Cycle 1 (28 days). The optimal dose of BKM120 was determined to be 60 mg by mouth (PO), once a day for each 28 day cycle along with bevacizumab, administered 10 mg/kg intravenously (IV) on Day 1 and Day 15 of each 28 day cycle.
Time Frame: Collected from day of first dose to the end of the first treatment cycle, up to 28 days
Population: Includes all Phase I patients receiving assigned study dosing.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I Dose Level 1 (60 mg BKM120, 10mg/kg Bevacizumab): Includes Phase I patients receiving 60 mg BKM120 and 10mg/kg bevacizumab.
- Phase I Dose Level 2 (80 mg BKM120, 10mg/kg Bevacizumab): Includes Phase I patients receiving 80mg BKM120 and 10mg/kg bevacizumab
Arm/Group | Phase I Dose Level 1 (60 mg BKM120, 10mg/kg Bevacizumab) | Phase I Dose Level 2 (80 mg BKM120, 10mg/kg Bevacizumab)
Number analyzed (Participants) | 6 | 6
Participants | 0 | 3

2. Primary Outcome: Median Progression-Free Survival (PFS) in Phase II Participants - Prior Bevacizumab and Bevacizumab Naive
Description: Two groups of patients in the Phase II trial will be considered separately, 1) participants who have not received previous bevacizumab and 2) participants who have received bevacizumab as part of first-line treatment. PFS is measured from the date of first protocol treatment until date of disease progression or death occurs, or date of last adequate tumor assessment using RANO or McDonald criteria. McDonald disease progression criteria: a 25% or greater increase in sum of the diameters of lesions, new lesions, or clinical deterioration (McDonald et al, 1990). RANO disease progression criteria: a 25% or greater increase in the enhancing lesions sum compared with smallest tumor measurement, significant increase in T2/FLAIR nonenhancing lesion on stable or increasing corticosteroids, new lesions, or clinical deterioration (Wen et al 2010)
Time Frame: every 8 weeks for up to 33 months
Population: All Phase II patients receiving at least one dose of study treatment that have had at least one post-baseline disease assessment
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase II Patients With Prior Bevacizumab Treatment.: Phase II patients previously treated with bevacizumab prior to enrolling in the study.
  Study treatment:
  BKM120: 60mg by mouth (PO), once a day for each 28 day cycle. Bevacizumab: 10 mg/kg administered intravenously (IV) on Day 1 and Day 15 of each 28 day cycle.
- Phase II Patients Without Prior Bevacizumab Treatment: Phase II patients that had not previously been treated with bevacizumab prior to enrolling in the study.
  Study treatment:
  BKM120: 60mg by mouth (PO), once a day for each 28 day cycle. Bevacizumab: 10 mg/kg administered intravenously (IV) on Day 1 and Day 15 of each 28 day cycle.
Arm/Group | Phase II Patients With Prior Bevacizumab Treatment. | Phase II Patients Without Prior Bevacizumab Treatment
Number analyzed (Participants) | 17 | 50
months | 2.8 [1.6 to 5.3] | 5.3 [3.6 to 9.2]

3. Secondary Outcome: Overall Response (CR or PR) of Phase II Participants - Prior Bevacizumab and Bevacizumab Naive
Description: Two groups of participants in the Phase II trial will be considered separately, 1) those who have not received previous bevacizumab and 2) those who have received bevacizumab as part of first-line treatment. Overall Response (OR) = number of patients with complete or partial responses (CR or PR) per McDonald or RANO criteria. McDonald: CR as disappearance of all disease for at least four weeks, no new lesions, no steroids; PR as 50% or greater decrease in the sum of all lesions compared with baseline for at least four weeks, no new lesions, stable or reduced steroids (McDonald 1990). RANO: CR as disappearance of all disease for at least 4 weeks, no new lesions, stable or improved nonenhancing lesions, and no steroid usage; and PR as a 50% or greater decrease in the sum of all lesions compared with baseline measurement for at least four weeks, no new lesions, stable or improved nonenhancing lesions on same or lower steroid dose compared to baseline (Wen 2010).
Time Frame: every 8 weeks, projected 24 months
Population: Includes participants in Phase II that receive at least one study treatment and have at least one post-baseline disease assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Phase II Participants - Prior Bevacizumab.: Phase II participants treated with bevacizumab as part of first-line treatment prior to enrolling in the study.
  Study treatment:
  BKM120: 60mg by mouth (PO), once a day for each 28 day cycle. Bevacizumab: 10 mg/kg administered intravenously (IV) on Day 1 and Day 15 of each 28 day cycle.
- Phase II Participants - Bevacizumab Naive: Phase II participants that have not received bevacizumab treatment prior to enrolling in the study.
  Study treatment:
  BKM120: 60mg by mouth (PO), once a day for each 28 day cycle. Bevacizumab: 10 mg/kg administered intravenously (IV) on Day 1 and Day 15 of each 28 day cycle.
Arm/Group | Phase II Participants - Prior Bevacizumab. | Phase II Participants - Bevacizumab Naive
Number analyzed (Participants) | 17 | 50
Participants | 1 | 18

4. Secondary Outcome: Median Overall Survival (OS) in Phase II Participants - Prior Bevacizumab and Bevacizumab Naive
Description: Two groups of patients in the Phase II trial will be considered separately, 1) participants who have not received previous bevacizumab and 2) participants who have received bevacizumab as part of first-line treatment. Overall survival is measured as the interval from first study treatment until date of death, or date last known alive.
Time Frame: every 12 weeks for up to 60 months
Population: Participants that have received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II Participants - Prior Bevacizumab | Phase II Participants - Bevacizumab Naive
Number analyzed (Participants) | 19 | 57
months | 6.6 [4.0 to 14.6] | 10.8 [9.2 to 13.5]

5. Secondary Outcome: Number of Participants With Grade 3/4/5 Serious Adverse Events and Adverse Events as a Measure of Safety and Tolerability
Description: Defined as the number of participants with treatment-emergent grade 3/4/5 adverse events/serious adverse events utilizing the National Cancer Institute Common Technology Criteria for Adverse Events (NCI CTCAE) v4.03
Time Frame: every 4 weeks for up to 5.2 years
Population: Includes all participants that received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Dose Level 1 (60 mg BKM, 10mg/kg Bevacizumab) | Phase I - Dose Level 2 (80 mg BKM120, 10mg/kg Bevacizumab) | Phase II - (60 mg BKM120, 10mg/kg Bevacizumab)
Number analyzed (Participants) | 6 | 6 | 76
Participants
  Fatigue | 1 | 0 | 8
  Confusion | 0 | 0 | 8
  Hyperglycemia | 1 | 0 | 5
  Diarrhea | 0 | 1 | 5
  Alanine aminotransferase increased | 0 | 1 | 5
  Hypertension | 0 | 0 | 6
  Seizure | 0 | 0 | 6
  Asthenia | 1 | 1 | 4
  Aspartate Aminotransferase Increased | 0 | 0 | 5
  Hypertriglyceridemia | 0 | 0 | 2
  Abdominal pain | 0 | 1 | 1
  Altered Mental Status | 0 | 1 | 1
  Gait Disturbance | 1 | 0 | 1
  Ataxia | 1 | 1 | 0
  Lipase Increased | 0 | 0 | 2
  Muscle Weakness | 0 | 0 | 2
  Pneumonia | 1 | 0 | 1
  Sepsis | 0 | 0 | 2
  Respiratory Failure | 1 | 0 | 1
  Thrombocytopenia | 0 | 0 | 1
  Hypercholesterolemia | 0 | 0 | 1
  Mucositis | 0 | 1 | 0
  Anorexia | 1 | 0 | 0
  Memory Impairment | 0 | 0 | 1
  Pruritis | 0 | 1 | 0
  Vomiting | 0 | 1 | 0
  Mood Alteration | 0 | 0 | 1
  Weight Loss | 0 | 0 | 1
  Neutropenia | 0 | 0 | 1
  Dehydration | 0 | 1 | 0
  Dyspnea | 0 | 0 | 1
  Hemorrhage | 0 | 0 | 1
  Somnolence | 1 | 0 | 0
  Taste Alteration | 0 | 1 | 0
  Agitation | 0 | 0 | 1
  Dysarthria | 0 | 0 | 1
  Fall | 0 | 0 | 1
  Hypermagnesemia | 0 | 0 | 1
  Ejection Fraction Decreased | 0 | 0 | 1
  Elevated Liver Enzymes | 0 | 0 | 1
  Hypoalbuminemia | 0 | 0 | 1
  Hypophosphatemia | 0 | 1 | 0
  Psychosis | 0 | 0 | 1
  Suicidal Ideation | 0 | 0 | 1
  Thromboembolic Event | 0 | 0 | 1
  Akathisia | 0 | 0 | 1
  Cellulitis | 1 | 0 | 1
  Chronic Obstructive Pulmonary Disease | 0 | 0 | 1
  Delirium | 1 | 0 | 0
  Diabetic Ketoacidosis | 0 | 0 | 1
  Enteritis | 0 | 1 | 0
  Female Genital Tract Fistula | 0 | 0 | 1
  Gastrointestinal Infection | 0 | 0 | 1
  Hyperlipidemia | 0 | 0 | 1
  Intracranial Hemorrhage | 0 | 0 | 1
  Left Ventricular Systolic Dysfunction | 0 | 0 | 1
  Necrotizing Fasciitis | 0 | 0 | 1
  Palsy | 0 | 0 | 1
  Paralysis | 0 | 0 | 1
  Personality Change | 0 | 0 | 1
  Syncope | 0 | 0 | 1
  Transaminitis | 0 | 0 | 1
  Urine Output Decreased | 0 | 0 | 1
  Vaginal Fistula | 0 | 0 | 1
  Volume Depletion | 0 | 1 | 0
  Headache | 0 | 1 | 2
  Hypokalemia | 0 | 0 | 4
  Hyponatremia | 0 | 0 | 3
  Nausea | 0 | 2 | 1
  Proteinuria | 0 | 0 | 3
  Rash | 0 | 1 | 2
  Urinary Tract Infection | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: Every 4 weeks up to 5.2 years
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were collected from day of first dose to 30 days after last dose of study medication and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Groups:
- Phase I - Dose Level 2 (80 mg BKM120, 10mg/kg Bevacizumab): BKM120: 60mg by mouth (PO), once a day for each 28 day cycle. Bevacizumab: 10 mg/kg administered intravenously (IV) on Day 1 and Day 15 of each 28 day cycle.
  Phase I patients include those diagnosed with advanced, metastatic solid tumors.
Arm/Group | Phase I - Dose Level 1 (60 mg BKM, 10mg/kg Bevacizumab) | Phase I - Dose Level 2 (80 mg BKM120, 10mg/kg Bevacizumab) | Phase II - (60 mg BKM120, 10mg/kg Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/6 | 27/76
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 75/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Dose Level 1 (60 mg BKM, 10mg/kg Bevacizumab) (N=6) | Phase I - Dose Level 2 (80 mg BKM120, 10mg/kg Bevacizumab) (N=6) | Phase II - (60 mg BKM120, 10mg/kg Bevacizumab) (N=76)
Seizure (Nervous system disorders) | 1 | 0 | 8
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0
Altered Mental Status (Nervous system disorders) | 0 | 1 | 1
Acute Ischemic Stroke (Nervous system disorders) | 0 | 0 | 1
Clostridium Difficile (Infections and infestations) | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Disease Progression (General disorders) | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Intracerebral Hemorrhage (Nervous system disorders) | 0 | 0 | 1
Intracranial Hemorrhage (Nervous system disorders) | 0 | 0 | 2
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Necrotizing Fasciitis (Infections and infestations) | 0 | 0 | 1
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rectovaginal Fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Upper GI Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Dose Level 1 (60 mg BKM, 10mg/kg Bevacizumab) (N=6) | Phase I - Dose Level 2 (80 mg BKM120, 10mg/kg Bevacizumab) (N=6) | Phase II - (60 mg BKM120, 10mg/kg Bevacizumab) (N=76)
Abdominal Pain (Gastrointestinal disorders) | 2 | 2 | 3
Abscess (Infections and infestations) | 1 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 2
Alanine Aminotransferase Increased (Investigations) | 2 | 1 | 26
Alkaline Phosphatase Increased (Investigations) | 1 | 0 | 3
Altered Mental Status (Psychiatric disorders) | 0 | 1 | 4
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 2 | 7
Anxiety (Psychiatric disorders) | 0 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 7
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 17
Asthenia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 10
Ataxia (Nervous system disorders) | 1 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6
Belching (Gastrointestinal disorders) | 1 | 2 | 0
Bloating (Gastrointestinal disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cerumen Impaction (Ear and labyrinth disorders) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 1 | 17
Constipation (Gastrointestinal disorders) | 1 | 0 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 6
Creatinine Levels Increased (Investigations) | 0 | 0 | 6
Cushingoid Facies (Endocrine disorders) | 1 | 0 | 0
Decreased Breath Sound (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Decreased Sensory Motor (Nervous system disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 2
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 10
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 18
Dizziness (Nervous system disorders) | 0 | 2 | 10
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Edema (General disorders) | 0 | 1 | 6
Elevated Liver Enzymes (Investigations) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Facial Pain (General disorders) | 1 | 0 | 0
Failure To Thrive (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 3 | 4 | 39
Gait Disturbance (General disorders) | 1 | 0 | 4
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 1 | 1
Hallucinations (Psychiatric disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 3 | 11
Hematuria (Renal and urinary disorders) | 0 | 1 | 3
Hemorrhage (Vascular disorders) | 2 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 0 | 4
Hypercholesterolemia (Metabolism and nutrition disorders) | 2 | 0 | 11
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 23
Hypersalivation (Gastrointestinal disorders) | 0 | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 16
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 8
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Infection (Infections and infestations) | 1 | 0 | 3
Insomnia (Nervous system disorders) | 1 | 0 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 10
Lipase Increased (Investigations) | 0 | 0 | 4
Memory Impairment (Nervous system disorders) | 0 | 2 | 7
Mood Alteration (Psychiatric disorders) | 0 | 3 | 5
Mucositis (Gastrointestinal disorders) | 0 | 1 | 11
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 4 | 13
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 7
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 5
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5
Palmar-Plantar Erythro (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Peripheral Neuropathy (Nervous system disorders) | 2 | 0 | 3
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 4 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 8
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 15
Rectal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 6
Skin Changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Skin Infection (Infections and infestations) | 1 | 1 | 0
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Somnolence (Nervous system disorders) | 1 | 0 | 3
Taste Alteration (Nervous system disorders) | 0 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 16
Thrush (Infections and infestations) | 1 | 0 | 1
Tooth Infection (Infections and infestations) | 1 | 0 | 1
Trace Protein Urinalysis (Investigations) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 3
Upper Respiratory Infection (Infections and infestations) | 2 | 0 | 8
Urinary Incontinence (Renal and urinary disorders) | 1 | 0 | 2
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 15
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 2
Vision Change (Eye disorders) | 0 | 1 | 1
Volume Depletion (Metabolism and nutrition disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 6
Weight Loss (Investigations) | 1 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites